CLINICAL TRIAL: NCT06154187
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel, Phase III Study to Evaluate the Efficacy and Safety of PBK_L2201 in Postmenopausal Women With Osteoporosis
Brief Title: Study to Evaluate the Efficacy and Safety of PBK_L2201 in Postmenopausal Women With Osteoporosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBK_L2201_301
Record Dates: First submitted 2023-11-20; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test 1 (Experimental): PBK_L2201
  Interventions: Drug: PBK_L2201
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBK_L2201 — Abaloparatide-SC 80 μg was to be self-administered daily using a Pen Injector device.
  Arms: test 1
Drug: Placebo — Placebo was formulated similar to abaloparatide-SC.
  Arms: placebo

SUMMARY:
This clinical trial was multicenter, randomized, double-blind, placebo-controlled, parallel, phase III bridge study.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy ambulatory postmenopausal woman from 50 to 85 years of age (inclusive) with osteoporosis.
* Be postmenopausal for at least 5 years. Postmenopausal status was established by a history of amenorrhea for at least 5 years and by an elevated serum follicle-stimulating hormone (FSH) value of ≥30 IU/L.
* Be to have a bone mineral density (BMD) T score ≤ -2.5 and > -5.0 at the lumbar spine or hip (femoral neck) by dual energy x-ray absorptiometry (DXA) and radiological evidence of 2 or more mild or one or more moderate lumbar or thoracic vertebral fractures, or history of low-trauma femoral, radius, humerus, sacral, pelvic, or ankle fracture within the past 5 years. Postmenopausal women older than 65 who meet the above fracture criteria but have a T score ≤ -2.0 and > -5.0 may be enrolled. Women older than 65 who do not meet the fracture criteria may also be enrolled if their T score is ≤ -3.0 and > -5.0

Exclusion Criteria:

* History of more than 4 spine fractures, mild or moderate, or any severe fractures.
* Presence of abnormalities of the lumbar spine that would prohibit assessment of spinal bone mineral density, defined as having at least 2 radiologically evaluable vertebrae within L1-L4.
* Unevaluable hip Bone mineral density (BMD) or patients who had undergone bilateral hip replacement (unilateral hip replacement was acceptable).

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density (BMD) change rate | 12 month
  The % change from baseline in lumbar spine Bone mineral density (BMD) through end of 12-month treatment.

SECONDARY OUTCOMES:
Bone mineral density (BMD) change | 12 month
  The change from baseline in lumbar spine Bone mineral density (BMD) through end of 12-month treatment.
Bone mineral density (BMD) change | 6 and 18 month
  The change & % change from baseline in lumbar spine Bone mineral density (BMD) through end of 6 and 18-month treatment.
Bone mineral density (BMD) % change | 6 and 18 month
  The change & % change from baseline in lumbar spine Bone mineral density (BMD) through end of 6 and 18-month treatment.
Bone mineral density (BMD) change | 6, 12 and 18 month
  The change & % change from baseline in total hip Bone mineral density (BMD) through end of 6, 12 and 18-month treatment.
Bone mineral density (BMD) % change | 6, 12 and 18 month
  The change & % change from baseline in total hip Bone mineral density (BMD) through end of 6, 12 and 18-month treatment.
Bone mineral density (BMD) change | 6, 12 and 18 month
  The change & % change from baseline in femoral neck Bone mineral density (BMD) through end of 6, 12 and 18-month treatment.
Bone mineral density (BMD) % change | 6, 12 and 18 month
  The change & % change from baseline in femoral neck Bone mineral density (BMD) through end of 6, 12 and 18-month treatment.
% incidence of new non-vertebral fractures | 12 month
  The % incidence of new non-vertebral fractures over 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Baek, Principal Investigator — The Catholic University of Korea Yeouido Saint Mary's Hospital
Locations (1):
- The Catholic University of Korea Yeouido Saint Mary's Hospital, Seoul, South Korea